CLINICAL TRIAL: NCT01454700
Title: The Effect of Sensor-Augmented Continuous Subcutaneous Insulin Infusion Compared to Multiple Daily Insulin Injections in Prevention of Increasing Urinary Albumin Excretion Rate in Type 1 Diabetes Mellitus
Brief Title: Effect of CSII and CGM on Progression of Late Diabetic Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steen Andersen (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Steen Andersen, Chief physician, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2011-122
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; Albuminuria; Late diabetes complications; CSII; CGM; Glycaemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Albuminuria | interventions — Insulin; Insulin Secretagogues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSII plus CGM (Experimental): Patients who has never been treated with insulin pump are randomized to 12 months with insulin pump therapy plus continuous glucose monitoring.
  Interventions: Device: Insulin pump therapy (CSII) plus continuous glucose monitoring (CGM)
- Multiple daily insulin injections (Active Comparator): randomized to 12 months standard/usual insulin regimen (multiple daily injections). (stays on insulin pen).
  Interventions: Other: Multiple daily insulin injections (MDI)

INTERVENTIONS:
Device: Insulin pump therapy (CSII) plus continuous glucose monitoring (CGM) — Randomization to 12 months with CSII plus CGM
  Other Names: CSII; CGM; Medtronic MiniMed Paradigm REAL-Time System; Medtronic MiniMed Paradigm Veo; Sensor augmented insulin pump therapy
  Arms: CSII plus CGM
Other: Multiple daily insulin injections (MDI) — Randomization12 months therapy with MDI
  Other Names: Human insulin; Insulin analogues
  Arms: Multiple daily insulin injections

SUMMARY:
The purpose of the study is to investigate whether the combination of insulin pump therapy and continued glucose monitoring (CGM) is superior to multiple daily insulin injections to prevent progression of albuminuria in patients with type 1 diabetes

DETAILED DESCRIPTION:
80 type 1 diabetic patients with kidney function (GFR > 45 ml/min), but with urine albumin excretion of at least 30 mg/day and HbA1c 7.5-13.0% are randomised to either multiple daily insulin injections (control group) or insulin pump therapy plus continued glucose monitoring (CGM) (intervention group). Patients must be in stable RAAS blockade before entering the study.

Before the study is initiated all patients receive education in intensive diabetes treatment and self-care including carbohydrate counting.

Patients return to the clinic after 1,3,6,9, and 12 months for measurement of urine albumine excretion, clinical examination including blood pressure, CGM sensor readings, four-point self monitored blood glucose (SMBG) profiles, blood samples and fulfillment of questionnaire to assess quality of life. At entry and after 12 months, eye fundus foto, 24-hour blood pressure, GFR, and carotis intima media thickness (CIMT)are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age,
* Type 1 diabetes according to WHO criteria,
* Urin albumine > 30 mg/g (albumine/creatinine ratio),
* HbA1c > 7.5 < 13.0%,
* No change in RAAS blocking treatment at least 4 weeks prior to screening.

Exclusion Criteria:

* Kidney disease other that diabetic nephropathy,
* Recurrence of severe hypoglycaemia or hypoglycaemia unawareness as judged by the investigator,
* Use of insulin pump within 12 months,
* Acute myocardial infarction within 3 months,
* Severe arteriosclerosis as judged by the investigator,
* Heart failure (NYHA class 3 or 4),
* Abuse of alcohol or drugs,
* Any cancer diagnosis unless in remission at least 5 years prior to screening,
* Participation in other intervention studies,
* Pregnant or lactating women,
* Any other disease, condition or type of treatment which - as judged by the investigator - render the patient ineligible to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
difference in change in urine albumine excretion from baseline to end of study (12 months) | 12 months
  Urine albumin excretion is evaluated at screening, at entry, after 1,3,6,9, and 12 months.

SECONDARY OUTCOMES:
difference in change of HbA1c from baseline to 12 months | 12 months
difference in change in self-monitored blood glucose (SMBG) measurement 4-point glucose profiles | 12 months
difference in change of 24-hour blood pressure | 12 months
difference in change of glomerular filtration rate (GFR) | 12 months
difference in the occurence or progression of retinopathy | 12 months
difference in change of cardiovascular biomarkers of inflammation, lipid metabolism and NT-proBNP | 12 months
difference in endothelial cell dysfunction | 12 months
difference in carotid intima media thickness (CIMT) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steen Andersen, MD, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Ranjan AG, Rosenlund SV, Hansen TW, Rossing P, Andersen S, Norgaard K. Improved Time in Range Over 1 Year Is Associated With Reduced Albuminuria in Individuals With Sensor-Augmented Insulin Pump-Treated Type 1 Diabetes. Diabetes Care. 2020 Nov;43(11):2882-2885. doi: 10.2337/dc20-0909. Epub 2020 Sep 4. PMID 32887707
- [Derived] Rosenlund S, Hansen TW, Rossing P, Andersen S. Effect of Sensor-Augmented Pump Treatment Versus Multiple Daily Injections on Albuminuria: A 1-Year Randomized Study. J Clin Endocrinol Metab. 2015 Nov;100(11):4181-8. doi: 10.1210/jc.2015-2839. Epub 2015 Sep 21. PMID 26390102